CLINICAL TRIAL: NCT07286006
Title: A Long-Term Extension Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 in Adult Patients With Graves' Disease
Brief Title: A Long-Term Extension Study of IMVT-1402 in Adult Participants With Graves' Disease (GD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMVT-1402-2505
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Graves' Disease
Keywords: IMVT-1402; Graves' disease; Immunoglobulin G; Thyroid-Stimulating Hormone Receptor; Antithyroid drug; FcRn
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: IMVT-1402
- Group B (No Intervention)
- Group C (No Intervention)

INTERVENTIONS:
Drug: IMVT-1402 — Dose 1 for up to 52 weeks
  Arms: Group A

SUMMARY:
This is a long-term extension study that will rollover participants completing feeder studies IMVT-1402-2502 (NCT06727604) or IMVT-1402-2503 (NCT07018323) to evaluate the efficacy and safety of IMVT-1402 in adult participants with GD. Eligible participants will be assigned to 1 of 3 study groups (Groups A, B and C) based on their GD status at the completion of their respective feeder study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed Study IMVT-1402-2502 or Study IMVT-1402-2503.
* Other, more specific inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have permanently discontinued IMP during the treatment period in the feeder study or have met study stopping criteria at any point up until the end of participation in the feeder study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Group A Participants who remain euthyroid, Off ATD, and Off IMVT-1402 | At Week 52

SECONDARY OUTCOMES:
Percentage of Group A Participants who are euthyroid and off ATD | At Week 26
Percentage of Group A Participants who are euthyroid and off ATD | Up to Week 52
Percentage of Group A Participants who are euthyroid, off ATD, and off IMVT-1402 | Up to Week 52
Time to earliest date of euthyroidism, off ATD, and off IMVT-1402 to the earliest date of confirmed relapse in Group A Participants | Up to Week 52
Percentage of Group B Participants who remain euthyroid, off ATD, and off IMVT-1402 | Up to Week 52
Percentage of Group B Participants who remain euthyroid, off ATD, and off IMVT-1402 | At Week 52
Time from Week 0 to the earliest date of confirmed relapse in Group B Participants | Up to Week 52
Percentage of Group C Participants who remain euthyroid, off ATD, and off IMVT-1402 | Up to Week 52
Percentage of Group C Participants who remain euthyroid, off ATD, and off IMVT-1402 | At Week 52
Time From Week 0 to the earliest date of confirmed relapse in Group C Participants | Up to Week 52
Percentage of Group A Participants who are euthyroid, off ATD, and seronegative for TRAb | At Week 26
Percentage of Group A Participants who are euthyroid, off ATD, and seronegative for TRAb | Up to Week 52

IPD SHARING:
Plan to Share IPD: No